CLINICAL TRIAL: NCT00698893
Title: An Open Study in Healthy Herpes Simplex Virus (HSV)-Positive Adults to Evaluate the Safety of GSK Biologicals' Candidate gD Vaccine, With or Without 3D MPL
Brief Title: Evaluation of Safety of Candidate gD Vaccine, With or Without MPL in Healthy Herpes Simplex Virus-positive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208141/001
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Herpes Simplex
Keywords: Herpes simplex; Herpes simplex candidate (gD) vaccine
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Herpes simplex candidate (gD) vaccine GSK208141
- Group B (Experimental)
  Interventions: Biological: Herpes simplex candidate (gD) vaccine GSK208141

INTERVENTIONS:
Biological: Herpes simplex candidate (gD) vaccine GSK208141 — Intramuscular injection, 2 doses, 2 different formulations (with and without MPL)

SUMMARY:
The purpose of the study is to evaluate the safety and reactogenicity of candidate gD vaccine, with or without MPL, in HSV-seropositive subjects. The immune response elicited in these subjects will also be evaluated.

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age
* Seropositive for antibodies against HSV
* Female volunteers must have been using contraceptives for at least 2 months before the entry and should avoid becoming pregnant for the duration of this study.
* Good physical condition as established by physical examination and history taking at the time of entry

Exclusion Criteria:

* Any abnormal laboratory value among the tests performed at screening.
* History of persistent hepatic, renal, cardiac or respiratory diseases
* Clinical signs of acute illness at the time of entry into the study.
* Previous history of asthma or hypersensitivity to drugs.
* Seropositive for antibodies against the human immunodeficiency virus
* Pregnancy and lactation.
* Treatment with corticosteroids or immunomodulating drugs.
* Simultaneous participation in another clinical trial.
* Administration of any other vaccine or immunoglobulins during the study period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 1992-05-01 (Actual); Primary Completion 1992-07-01 (Actual); Study Completion 1992-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the vaccine safety by repeated physical examination and by recording all local and general signs/symptoms | Throughout the study
Measurement of haematology/biochemical parameters on blood samples | Throughout the study
Vaccine reactogenicity by soliciting of local and general signs/symptoms | On the day of vaccination and the subsequent 7 days
Vaccine immunogenicity by 6 measurements of anti-HSV antibodies | From day 0 to day 45 following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Results for study 208141/001 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/208141/001?search=study&#rs